CLINICAL TRIAL: NCT03705351
Title: Safety and Tolerability of Tumor Treating Fields (TTFields) Combined With Chemoradiation in Newly Diagnosed Glioblastoma (Unity)
Brief Title: Tumor Treating Fields With Chemoradiation in Newly Diagnosed GBM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Prinicipal Investigator departure from institution
Sponsor: Providence Health & Services (Other)
Collaborators: University of California, San Francisco (Other); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UNITYGBM01
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-08

CONDITIONS: Glioblastoma; Cancer of Brain; Glioblastoma Multiforme; Brain Tumor
Keywords: temozolomide; tumor treating fields; optune; novocure; glioblastoma; brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: The study is an open-label pilot study. Following surgery, eligible patients will start tumor treating fields therapy with the Optune device less than 2 weeks prior to radiation and temozolomide given at a dose and schedule conforming to routine treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Patients will receive trimodal therapy consisting of tumor treating fields therapy with the Optune device concurrent with temozolomide and radiation therapy.
  Interventions: Device: Tumor Treating Fields; Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Device: Tumor Treating Fields — Optune is intended as a treatment for adult patients (22 years of age or older) with histologically-confirmed glioblastoma multiforme (GBM). Treatment will begin approximately 1 week prior to start of radiation and temozolomide treatment and continue concurrently throughout the duration of the study.
  Other Names: Optune; Novocure
Drug: Temozolomide — Patients will be given temozolomide according to routine treatment dosing and schedule.
  Other Names: Temodar
Radiation: Radiation Therapy — Patients will be given radiation therapy according to routine treatment dosing and schedule.

SUMMARY:
The study is an open-label pilot study in newly diagnosed glioblastoma patients following surgery. Eligible patients will receive treatment with tumor treating fields therapy using the Optune device starting less than 2 weeks prior to start of chemoradiation. Patients will receive radiation and temozolomide at a routine treatment dose and schedule.

DETAILED DESCRIPTION:
The study is an open-label pilot study in newly diagnosed glioblastoma patients following surgery. Eligible patients will receive treatment with tumor treating fields therapy using the Optune device starting less than 2 weeks prior to start of chemoradiation. Patients will receive radiation and temozolomide at a routine treatment dose and schedule.

The expected toxicity is skin related, and patients will be followed closely with weekly skin and neurological examinations during radiation therapy and for 8 weeks afterwards to capture any delayed toxicity as they begin adjuvant therapy per routine treatment. As long as study treatment is tolerated and their conditions remain stable, patients will continue the treatment for up to 24 months.

Prior to enrollment, an exploratory analysis of radiation dosimetry will be performed by phantom modeling incorporating the Optune arrays. The study incorporates three stages of recruitment to confirm the safety of combining tumor treating fields therapy with concurrent chemoradiation: a safety lead-in cohort of the first 6 patients enrolled, a second safety lead-in cohort of 9 patients, and an expansion cohort with 15 additional patients.

ELIGIBILITY:
Inclusion Criteria:

1. GBM or Gliosarcoma by histology
2. MGMT methylation status and IDH mutation status must be assessed at the study site or patient's referral center. MGMT status will be used for stratification purposes but will not exclude patients from this study if they are either methylated, unmethylated, or indeterminate, or in process at the time of enrollment. Similarly, subjects with tumors that are IDH mutated or wild type are both eligible.
3. Supratentorial location
4. Maximum safe resection (including patients who can only safely be biopsied)
5. 22 years of age or older
6. Estimated survival of at least 12 weeks
7. KPS 70% or greater at time of entry to study
8. Patient provided written informed consent, or provided by a legally authorized representative
9. Willingness to comply with all procedures, including visits or evaluations, imaging, laboratory tests and rescue measures
10. Acceptable method of birth control (see appendix)
11. Have had a contrast-enhanced brain MRI after tumor resection procedure. If biopsy alone performed, cranial CT may be used in place of MRI, only if the patient had a preoperative MRI scan within 14 days of the biopsy.
12. The following time period must have elapsed prior to study enrollment: 3-6 weeks (21-42 days) from time of definitive surgery or 2-4 weeks (14-28 days) from the time of biopsy, for those who were only able to safely have a biopsy and not full resection.

Exclusion Criteria:

1. Craniotomy or stereotactic biopsy wound dehiscence or infection
2. Known by history to be HIV positive or to have an AIDS-related illness, active Hepatitis B, or active Hepatitis C (testing not required)
3. Presence of skull defects (bullets, metal fragments, missing bone)
4. Patients with implanted electronic medical devices (including but not limited to: pacemaker, vagal nerve stimulator, or pain stimulator)
5. Prior invasive malignancy, unless disease free for 3 or more years, with the exception of basal cell carcinoma, cervical carcinoma in situ, or melanoma in situ
6. Recurrent malignant gliomas or higher grade gliomas transformed from previous low grade (II) glioma
7. Patients with any current Primary brain stem or spinal cord tumor
8. Prior use of temozolomide
9. Prior treatment with Avastin
10. Individuals requiring >8mg of dexamethasone per day within 7 days prior to Day 1 (high dose steroid taper following craniotomy with >8mg of dexamethasone is allowed during the screening period, but subjects must taper down to 8mg or less of dexamethasone (or bioequivalent) within 7 days prior to Day 1).
11. Clinically significant lab abnormalities at screening showing bone marrow, hepatic, and renal dysfunction:

    * Thrombocytopenia (platelet count < 100 x 103/μL)
    * Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
    * Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
    * Total bilirubin > upper limit of normal
    * Significant renal impairment (serum creatinine > 1.7 mg/dL)
12. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting) at screening
13. Inability to swallow pills
14. Clinically significant or unstable comorbid medical condition, per investigator discretion (for example, active or uncontrolled infection requiring systemic therapy, including known HIV or hepatitis B or C virus)
15. Known current alcohol or drug abuse, per investigator discretion. Prior history of substance abuse is permissible if subject has been sober for the past 3 years.
16. Any clinically significant psychiatric condition that would prohibit patient willingness or ability to successfully complete study procedures, per investigator discretion
17. Patients with an allergy to or an inability to have gadolinium contrast dye administered with MRI
18. Patients with aneurysm clips or implanted metal objects in the brain
19. Patients with significant skin breakdown on the scalp
20. Patients who cannot receive standard of care radiation therapy and can only receive hypofractionated radiation due to age and poor performance status , per investigator discretion

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Chen, MD, Principal Investigator — Providence Health and Services
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Providence St. Vincent Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Brain & Spine Institute Clinical Research — https://oregon.providence.org/our-services/c/clinical-trials-brain/

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety lead-in Cohort: Participants who finished the DLT period and were assessed by investigators
Period: Overall Study
Arm/Group | Safety lead-in Cohort
Started | 7
Completed | 0
Not Completed | 7
Not completed — Study termination | 3
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Newly diagnosed patients histologically confirmed glioblastoma after maximally safe resection
Arm/Group | Safety lead-in Cohort
Number analyzed (Participants) | 7
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57 [47.50 to 63.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Karnofsky Performance Scale (KPS) [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses.
  Participants
    KPS 70: Cares for self; unable to carry on normal activity or to do active work | 1
    KPS 80: Normal activity with effort; some signs or symptoms of disease | 3
    KPS 90: Able to carry on normal activity, minor signs or symptoms of disease | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treatment-Related Adverse Events Associated With Trimodal Therapy
Description: Number of patients who experienced a treatment-related adverse event
Time Frame: 15 Weeks (8 weeks after completion of trimodal therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety lead-in Cohort
Number analyzed (Participants) | 7
Participants | 2

2. Primary Outcome: Severity of Treatment-Related Adverse Events Associated With Trimodal Therapy
Description: Number of patients who experienced a treatment-related serious adverse event based on the NCI Common Terminology Criteria for Adverse Events (version 4.03)
Time Frame: 15 weeks (8 weeks after completion of trimodal therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety lead-in Cohort
Number analyzed (Participants) | 7
Participants | 2

3. Secondary Outcome: Overall Survival Rate
Description: Number of patients alive at Day 106 (15 weeks), end of main study period
Time Frame: Day 106
Measure: Count of Participants; unit: Participants
Arm/Group | Safety lead-in Cohort
Number analyzed (Participants) | 7
Participants
  Number of participants alive at Day 106 | 5
  Number of participants not evaluated due to being withdrawn from study prior to Day 106 | 2

4. Secondary Outcome: Progression-free Survival at 6 Months and 24 Months
Description: Number of patients who are progression free at 6 months and 24 months. Progression is defined as any of the following: greater than or equal to 25% increase in sum of lesions compared with smallest tumor measurement obtained, significant increase in T2/FLAIR non-enhancing lesions, any new lesion, clear clinical deterioration not attributable to other causes, or clear progression of non-measureable disease.
Time Frame: 6 months and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety lead-in Cohort
Number analyzed (Participants) | 7
Participants
  Number of participants progression-free at 6 months | 3
  Number of participants progression-free at 24 months | NA — Study terminated prior to any patient reaching Month 24

ADVERSE EVENTS:
Time Frame: 15 weeks (8 weeks after completion of trimodal therapy)
Arm/Group | Safety lead-in Cohort
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety lead-in Cohort (N=7)
Thrombocytopenia - worsened (Blood and lymphatic system disorders) | 1 (1)
Decreased lymphocytopenia (Investigations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety lead-in Cohort (N=7)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anemia (decreased hemoglobin) (Blood and lymphatic system disorders) | 1 (1)
Pain in lymph node, right cervical region (Blood and lymphatic system disorders) | 1 (1)
Enlarged lymph node right cervical region (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia - worsened (Blood and lymphatic system disorders) | 1 (1)
Eye strain - right eye (Eye disorders) | 1 (1)
Right Field Cut (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Mild constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Nausea - worsened from baseline (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Fatigue in evenings (General disorders) | 1 (1)
Generalized fatigue (General disorders) | 3 (3)
Impaired tandem gait (General disorders) | 1 (1)
Allergic reaction due to OPTUNE - rash - diffuse (Immune system disorders) | 1 (1)
Allergic reaction - rash, diffuse unknown origin (Immune system disorders) | 1 (1)
Itching due to allergic reaction - diffuse, unknown origin (Immune system disorders) | 1 (1)
Conjunctivitis in left eye (Infections and infestations) | 1 (1)
Bruising on abdomen, secondary to itching (Injury, poisoning and procedural complications) | 1 (1)
Scabs on knees from falls (Injury, poisoning and procedural complications) | 1 (1)
Increased ALT (Investigations) | 1 (1)
Increased creatinine (Investigations) | 1 (1)
Increased glucose (Investigations) | 1 (1)
Decreased albumin (Investigations) | 1 (1)
Decreased calcium (Investigations) | 1 (1)
Decreased lymphocytes (Investigations) | 1 (3)
Lymphocytes, decreased (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Slight weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dull, throbbing headached - lower right side back of head (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 2 (2)
Facial Muscle Weakness (Left Side) (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Headaches - intermittent (Nervous system disorders) | 1 (1)
Headache - worsened from baseline (Nervous system disorders) | 1 (1)
Imbalance (Nervous system disorders) | 1 (1)
Left sided weakness (Nervous system disorders) | 1 (3)
Memory Impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Tingling - right side of face (Nervous system disorders) | 1 (1)
Tingling in fingers - both hands (Nervous system disorders) | 1 (1)
Twitch on top of head - intermittent (Nervous system disorders) | 1 (1)
Worsening Imbalance (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blisters on scalp - diffuse (Skin and subcutaneous tissue disorders) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin on scalp - front left side (Skin and subcutaneous tissue disorders) | 1 (1)
Dryness of skin on scalp - diffuse (Skin and subcutaneous tissue disorders) | 1 (1)
Dryness on scalp - diffuse (Skin and subcutaneous tissue disorders) | 1 (1)
Edema - scalp - right side (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema, scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema of temples (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema on scalp - front left side (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema scalp - circumferential under diodes (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema scalp - diffuse (Skin and subcutaneous tissue disorders) | 2 (2)
Folliculitis - back of hand (Skin and subcutaneous tissue disorders) | 1 (1)
Folliculitis on lower back of head (Skin and subcutaneous tissue disorders) | 1 (1)
Itching on scalp - diffuse (Skin and subcutaneous tissue disorders) | 1 (2)
Itchy scalp - location not specified (Skin and subcutaneous tissue disorders) | 1 (1)
Moist dsequamation - right side of head (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp blisters - diffuse (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp peeling - left frontal lobe (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Three open sores on front left side of scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Two blisters on the back of head (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03705351/Prot_SAP_000.pdf